CLINICAL TRIAL: NCT07085598
Title: Effect of Vitamin D3 Supplementation on Cardiac Autonomic Nerve Function in Male Epileptic Patients With Hypovitaminosis D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bangladesh Medical University (Other)
Responsible Party: Principal Investigator, Samikha Sarker, Principal Investigator, Bangladesh Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 5592
Record Dates: First submitted 2025-07-12; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Epilepsy
Keywords: Vitamin D3; Hypovitaminosis D; HRV
MeSH Terms: conditions — Epilepsy; Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Intervention Model Description: 15 epileptic patients with hypovitaminosis D will be enrolled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 15 male epileptic patients with hypovitaminosis D (Experimental): 15 male epileptic patients with hypovitaminosis D will be enrolled. They will be supplemented with Vitamin D orally 50,000 IU/week for 8 weeks
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Vitamin D — 15 male epileptic patients with hypovitaminosis D will be enrolled. They will be supplemented with Vitamin D orally 50,000 IU/week for 8 weeks

SUMMARY:
The goal of this clinical trial is to see the effect of vitamin D3 supplementation on cardiac autonomic nerve function in male epileptic patients with hypovitaminosis D that weather vitamin D improves heart rate variability or not. The main questions it aims to answer are:

1. Does vitamin D improves cardiac autonomic tone in male epileptic patients?
2. Does vitamin D improves heart rate variability in male epileptic patients?

It is a self control trial. Participants will:

1. undergo through baseline HRV testing
2. start to take vitamin D3 50000 IU once in a week for 8 weeks

b) visit the university after 8 weeks for post interventional HRV testing . Researcher will compare the pre test and post test value of HRV testing.

DETAILED DESCRIPTION:
In epilepsy, there is a shifting of autonomic balance toward sympathetic dominance & heart rate variability (HRV) is reduced which can be detected by interictal heart rate variability (HRV) testing. Patients treated with anti-epileptic drugs (AEDs) are suffered from one of its major adverse effects of vitamin D3 deficiency or hypovitaminosis D due to enzyme inducing effect of AEDs. Vitamin D3 is a neuroprotective hormone that modulates autonomic balance and regulates sympathetic and parasympathetic nervous systems. Vitamin D3 deficiency is also associated with the risk of reduced HRV. Administration of vitamin D3 in vitamin D3 deficient epileptic patients may improve their cardiac autonomic nerve function that can be interpreted by HRV.

ELIGIBILITY:
Inclusion Criteria:

* • Diagnosed male patients with Epilepsy by neurologist from the OPD of Department of Neurology by taking proper history of at least two unprovoked (or reflex) seizures occuring > 24 hours apart, from patients and eye witnesses.

  * Having hypovitaminosis D (serum vitamin D3 level <30 ng/ml)
  * Age: 20-40 years.

    * Sex: Male
    * BMI : 18.5-24.9 kg/m2
    * Taking antiepileptic drug for 6 months to 2 years ( Enzyme inducer AEDs, e.g. Carbamazepine, Phenytoin, Phenobarbital)
    * Without medication that affect central nervous system other than antiepileptic drugs (AEDs).

Exclusion Criteria:

* • Epileptic patients taking Sodium valproate, oxcarbazepine, Topiramate, Lamotrigine, Levetiracetam.

  * Patient having absence seizure
  * Alcoholic
  * Smoker
  * Patients taking following drugs will be excluded-

    * Anti-diabetic drugs
    * Antioxidant vitamin supplements
    * Antihypertensive drug
    * Anti-arrhythmic drug
    * Lipid lowering medications
    * Sedatives
  * Patients having known hypersensitivity to vitamin D3
  * All patients with the history of or currently suffering from following diseases & condition will be excluded-

    * Cardiovascular disorders (Myocardial infarction, coronary heart disease, cardiac arrhythmia, CCF)
    * Other neurological disorders (Migraine, stroke)
    * Respiratory disorders (Bronchial asthma, COPD)
    * Renal insufficiency (S. Creatinine > 1.5 mg/dl, Acute or chronic kidney disease)
    * Endocrine disease (Diabetes mellitus, Thyroid disorders- hypothyroidism, hyperthyroidism)
    * Arthritis (rheumatoid arthritis)
    * Liver diseases
    * Neoplastic disease
    * Psychiatric disorder (schizophrenia, bipolar disorder)
    * Current use of iron, zinc, calcium, magnesium and multivitamin supplementation
    * Already performing yoga or breathing exercise
    * Patients with hypercalcemia

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Vitamin D3 supplementation has effects on cardiac autonomic nerve function in male epileptic patients with hypovitaminosis D. | 8 weeks
  In epilepsy, cardiac autonomic nerve function is altered which can be measured by heart rate variability test(HRV). HRV is reduced in epilepsy. Vitamin D3 supplementation in patients with epilepsy will improve their cardiac autonomic nerve function which can be detected by measuring various parameters of HRV test such as SDRR, LF(Low frequency).

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Samikha Sarker, MBBS, MD Resident (Phase B), Principal Investigator — BMU
Locations (1):
- Bangladesh Medical University, Dhaka, Shahbag, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Teagarden DL, Meador KJ, Loring DW. Low vitamin D levels are common in patients with epilepsy. Epilepsy Res. 2014 Oct;108(8):1352-6. doi: 10.1016/j.eplepsyres.2014.06.008. Epub 2014 Jul 6. PMID 25060996